CLINICAL TRIAL: NCT00769236
Title: Evaluation of Intestinal Secretion of Antibodies and Auto-antibodies Associated With Crohn's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2008-A00080-55; 2008-05
Record Dates: First submitted 2008-10-08; First posted 2008-10-09 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Crohn's Disease
MeSH Terms: conditions — Crohn Disease | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Other): Patients with crohn disease
  Interventions: Other: Blood sampling and biopsy
- 2 (Other): Patients reached by hemorrhagic first side-colitis
  Interventions: Other: Biopsy and blood sampling
- 3 (Other): Patients controls
  Interventions: Other: Biopsy and blood sampling

INTERVENTIONS:
Other: Blood sampling and biopsy — Biopsy and blood : Research for various antibodies
  Arms: 1
Other: Biopsy and blood sampling — Biopsy and blood : research for various antibodies
  Arms: 2
Other: Biopsy and blood sampling — Blood and biopsy : research for various antibodies
  Arms: 3

SUMMARY:
We propose to study the intestinal secretion of ASCA by evaluating them in biopsy culture supernatants from a cohort of patients suffering from CD (n=80) and a cohort of control patients (UC (n=40) and patients without IBD (n=40 )).

DETAILED DESCRIPTION:
Its diagnosis is based upon clinical, endoscopic and histological parameters but recent studies have shown that seric evaluation of immunological markers (anti-Saccharomyces cerevisiae antibodies (ASCA), anti-neutrophil cytoplasmic auti-antibodies (ANCA)) could be useful. Crohn's disease (CD) is an inflammatory bowel disease (IBD) of the young people. Antibodies anti-chitobisoside carbohydrate (ACCA), anti-laminaribioside carbohydrate (ALCA) and anti-mannobioside carbohydrate (AMCA) have been described as new serological markers of CD.

ELIGIBILITY:
Inclusion Criteria:

* Patients reached by disease of crohn
* patients reached by hemorrhagic first side-colitis

Exclusion Criteria:

* Forms ileales or ano-périneales pure of disease of crohn
* indefinite colitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2008-06; Primary Completion 2010-05 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Compare the performances of the dosage of the ASCA in floating it of culture of intestinal biopsies in that of their dosage in the serum | 24 months

SECONDARY OUTCOMES:
Determine if the patients reached by disease of crohn not presenting ASCA in their serum represent one under group of disease of crohn | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Sophie Desplat-Jego, MD, Principal Investigator — Assistance Publique des Hopitaux de Marseille
Locations (1):
- Laboratoire d'Immunologie - Hopital de la Conception, Marseille, France